CLINICAL TRIAL: NCT00797134
Title: Retinal Thickness Analysis Using Optical Coherence Tomography
Status: Completed | Type: Observational
Sponsor: Association for Innovation and Biomedical Research on Light and Image (Other)
Responsible Party: Sponsor
Other Study IDs: CNTM025AOCT
Record Dates: First submitted 2008-11-24; First posted 2008-11-25 (Estimated); Last update posted 2015-02-03 (Estimated); Status verified 2015-02

CONDITIONS: Diabetic Retinopathy
MeSH Terms: conditions — Diabetic Retinopathy

STUDY DESIGN:
Observational Model: Cohort
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- DR: Diabetic Retinopathy

SUMMARY:
The main objective of this study is to characterize and correlate diabetic macular edema (DME), i.e. increased retinal thickness, measured by Optical Coherence Tomograph (OCT), and retinal visual function.

The secondary objectives of this study are the analysis and characterization of DME progression over time (between two visits), and the comparison of OCT data obtained with different devices.

The results of this study will be used exclusively for scientific purposes.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of DR
* Females or Males
* Age over 18 years
* Signed Informed Consent Form

Exclusion Criteria:

* Cataract or other eye disease that may interfere with fundus examinations
* Vitreous syneresis or posterior vitreous detachment
* Dilatation of the pupil < 5 mm

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects followed regularly by their ophthalmologist performing, as part of their follow-up, optical coherence tomography with OCT, and fulfilling the inclusion/exclusion criteria will be included.
Sampling Method: Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2008-11; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Retinal thickness. | After visit(s)

SECONDARY OUTCOMES:
Choroidal Thickness | After visit(s)

CONTACTS AND LOCATIONS:
Overall Officials: José Cunha-Vaz, MD, PhD, Principal Investigator — Association for Innovation and Biomedical Research on Light and Image
Locations (1):
- AIBILI, Coimbra, Coimbra District, Portugal

REFERENCES:
- See also: Related Info — http://www.aibili.pt